CLINICAL TRIAL: NCT00556959
Title: A Phase III, Dose-Response Evaluation of the Efficacy and Safety of CLONICEL® (Clonidine HCl Sustained Release) vs. Placebo in the Treatment of Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Study Evaluating the Safety and Efficacy of CLONICEL® to Treat Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Addrenex Pharmaceuticals, Inc. (Industry)
Responsible Party: Moise Khayrallah, PhD / President & CEO, Addrenex Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLON-301
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2010-03-24 (Estimated); Status verified 2008-08

CONDITIONS: Attention Deficit Disorder With Hyperactivity
Keywords: ADHD; Clonidine; Attention Deficit; Hyperactivity; CLONICEL; Addrenex
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Spasm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): CLONICEL High Dose
  Interventions: Drug: high dose clonidine HCl sustained release
- 2 (Experimental): CLONICEL Low Dose
  Interventions: Drug: low dose clonidine HCl sustained release
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: high dose clonidine HCl sustained release — high dose clonidine HCl sustained release tablets for 8 weeks
  Arms: 1
Drug: low dose clonidine HCl sustained release — low dose clonidine HCl sustained release tablets for 8 weeks
  Arms: 2
Drug: placebo — placebo tablets for 8 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to determine whether CLONICEL® (clonidine HCl sustained release) is a safe and effective treatment for children and adolescents with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
Clonidine is a centrally acting alpha2 adrenergic agonist that has been used effectively since the early 70s to treat mild to moderate hypertension. In addition to hypertension, clonidine has been evaluated and used extensively for several other indications, including attention deficit hyperactivity disorder (ADHD).

An easy to administer clonidine formulation is needed that retains the efficacy of the current oral formulation but has an improved safety profile. The current trial will investigate the safety and efficacy of clonidine delivered from the sustained release formulation of CLONICEL in the treatment of children and adolescents with ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 6 and 17 years of age, inclusive
* Diagnosis of ADHD of the hyperactive or combined inattentive/hyperactive subtypes according to DSM-IV criteria
* Minimum score of 26 on the ADHDRS-IV questionnaire at Baseline
* General good health as judged by the Principal Investigator
* Body mass index ≥ 5th percentile of the subject's age group according to the CDC growth chart.
* Ability to swallow tablets
* General IQ ≥80 as judged by the Principal Investigator
* Subject as well as parent/guardian able to sign informed assent or consent form.

Exclusion Criteria:

* If female of child-bearing potential, pregnant or lactating or does not agree to use a medically acceptable form of birth control, such as hormonal medication, double-barrier method, or IUD
* Presence of a clinically significant illness or abnormality on physical examination or clinical laboratory evaluations that, in the opinion of the investigator, would increase the safety risks from clonidine administration or interfere with the ability of the patient to take part in the study.
* Presence of clinically significant abnormality on centrally interpreted Electrocardiogram (ECG) readings
* History or presence of a concomitant psychiatric disorder requiring psychotropic medication or a severe concomitant Axis I or Axis II disorder that could interfere with study assessments in the judgment of the Principal Investigator
* History of concomitant conduct disorder (CD)
* History of seizures, except for a single episode of febrile seizure prior to age 2
* History of syncopal episodes
* Presence of a disorder that would interfere with the absorption, metabolism, or excretion of clonidine
* History of intolerance to clonidine, including any dermatologic reaction to transdermal clonidine
* Presence or history of alcohol or drug abuse
* Positive drug screen, with the exception of ADHD drugs
* Use of any investigational drug within 30 days of study start.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 236 (Actual)
Dates: Start 2007-10; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
ADHDRS-IV | Week 5

SECONDARY OUTCOMES:
CPRS-L, CGI-S, and CGI-I | Week 5
Adverse Events, Laboratory Assessments, Vital Signs, and ECGs | Throughout Treatment Phase

CONTACTS AND LOCATIONS:
Overall Officials: Moise A Khayrallah, PhD, Study Director — Addrenex Pharmaceuticals, Inc.
Locations (12):
- United States (12):
  - Gainesville, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Rochester Hills, Michigan
  - Clementon, New Jersey
  - Voorhees Township, New Jersey
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Oklahoma City, Oklahoma
  - Houston, Texas
  - Lake Jackson, Texas

REFERENCES:
- [Derived] Jain R, Segal S, Kollins SH, Khayrallah M. Clonidine extended-release tablets for pediatric patients with attention-deficit/hyperactivity disorder. J Am Acad Child Adolesc Psychiatry. 2011 Feb;50(2):171-9. doi: 10.1016/j.jaac.2010.11.005. PMID 21241954